CLINICAL TRIAL: NCT03381664
Title: A Phase 1, Randomized, Single-Dose, 3-Way, Crossover Study to Compare the Relative Bioavailability, Pharmacokinetics, Safety and Tolerability of AVP-923 (Dextromethorphan Hydrobromide and Quinidine Sulfate Capsules) Administered in Applesauce or Via a Nasogastric Feeding Tube With Administration of a Capsule in Healthy Adult Subjects
Brief Title: Study to Assess the Bioavailability, Pharmacokinetics, Safety, and Tolerability of AVP-923 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-AVR-135
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: bioavailability; pharmacokinetics; safety; tolerability; AVP-923; dextromethorphan; quinidine
MeSH Terms: interventions — dextromethorphan - quinidine combination; Dextromethorphan; Quinidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AVP-923-20/10 capsule (Experimental): Participants will receive a single AVP-923-20/10 (dextromethorphan hydrobromide [DM] 20 milligram [mg]/quinidine sulfate [Q] 10 mg) capsule administered orally.
  Interventions: Drug: AVP-923
- AVP-923-20/10 via applesauce (Experimental): Participants will receive the contents from a single AVP-923-20/10 capsule mixed and consumed in 1 tablespoon of applesauce.
  Interventions: Drug: AVP-923
- AVP-923-20/10 via nasogastric feeding tube (Experimental): Participants will receive the contents from a single AVP-923-20/10 capsule solubilized in feeding solution and administered through a nasogastric feeding tube.
  Interventions: Drug: AVP-923

INTERVENTIONS:
Drug: AVP-923 — capsule
  Other Names: Dextromethorphan Hydrobromide and Quinidine Sulfate

SUMMARY:
This study will be conducted to evaluate the relative bioavailability, pharmacokinetics, safety, and tolerability of AVP-923 (dextromethorphan hydrobromide [DM] and quinidine sulfate [Q] capsules) when the contents of a capsule are administered in applesauce or via a nasogastric feeding tube, compared with administration of a capsule in healthy, fasting, adult participants.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized, single-dose, 3-treatment, 3-period, 6-sequence crossover study in healthy adult participants consisting of approximately 7 weeks of treatment. The study population will be limited to extensive metabolizers of cytochrome P450 (CYP) 2D6.

Approximately 18 participants will be randomly assigned to 1 of 6 sequences (ABC, ACB, BAC, BCA, CAB, CBA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, 18 to 65 years of age, inclusive
* Willing to sign informed consent form
* Cytochrome P450 2D6 genotype that confers extensive metabolizer profile (as per documented phenotype interpretation from local laboratory and approval from Avanir)

Exclusion Criteria:

* History or presence of significant pulmonary, hepatic, renal, hematologic, allergic, endocrine (including diabetes), immunologic, dermatologic, neurologic (including history or presence of seizures or convulsive disorders), psychiatric disease (including history of suicidal ideation or behavior) or any eating disorder deemed clinically significant by the investigator
* History or presence of significant cardiovascular disease, including complete heart block, QT interval corrected for heart rate (QTc) prolongation, and/or torsades de pointes
* History or presence of any gastrointestinal (GI) disease or condition that could compromise participant safety or affect the absorption of study drug, including GI ulcers, GI bleeding, esophageal or gastric varices, and dyspepsia requiring regular (i.e., more frequently than once a month) use of acid-reducing drugs
* Known hypersensitivity/intolerance to dextromethorphan or quinidine
* Participants whom the principal investigator or his delegate deems to be ineligible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Mean area under the concentration time curve (AUC) from time 0 to time of last measurable concentration (AUC0-t) for the analytes dextromethorphan (DM), dextrorphan (DX), 3-methoxymorphinan (3-MM), and quinidine (Q) | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)
Mean AUC from time 0 to infinity (AUC0-inf) for the analytes DM, DX, 3-MM, and Q | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)
Mean maximum plasma concentration (Cmax) for the analytes DM, DX, 3-MM, and Q | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)
Mean time to maximum plasma concentration (Tmax) for the analytes DM, DX, 3-MM, and Q | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)
Mean apparent terminal elimination half-life (t1/2) for the analytes DM, DX, 3-MM, and Q | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)
Mean apparent elimination rate constant (kel) for the analytes DM, DX, 3-MM, and Q | pre-dose (within 30 minutes prior to dosing) and post-dose (up to 48 hours after drug administration)

SECONDARY OUTCOMES:
Number of participants with any adverse event | 3 weeks
Number of participants with any clinically significant clinical laboratory evaluation | 3 weeks
  Clinical significance will be determined by the Investigator.
Number of participants with any clinically significant physical examination evaluation | 3 weeks
  Clinical significance will be determined by the Investigator.
Number of participants with any clinically significant electrocardiogram evaluation | 3 weeks
  Clinical significance will be determined by the Investigator.
Number of participants with any clinically significant vital sign value | 3 weeks
  Clinical significance will be determined by the Investigator.
Number of participants with the indicated score on the Columbia-Suicide Severity Rating Scale (C-SSRS) | 3 weeks
  The C-SSRS will be used to prospectively assess suicidal ideation (intensity rated from 1 [low severity] to 5 [high severity]) and behavior throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States